CLINICAL TRIAL: NCT06495255
Title: Bioavailability of Human Milk Oligosaccharides in Healthy Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bonn (Other)
Collaborators: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Marie-Christine Simon, PhD MSc RD, Jun. Prof. Dr. Marie-Christine Simon (PI), University of Bonn
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 299/22
Record Dates: First submitted 2024-05-14; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Healthy
Keywords: absorption; excretion; metabolic markers

STUDY DESIGN:
Intervention Model Description: Two or more interventions, each alone and in combination, are evaluated in parallel
Who Masked: Participant
Masking Description: Participants are blinded to the supplement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): HMO bolus administration
  Interventions: Dietary Supplement: Human Milk Oligosaccharides (HMOs)
- Control (Experimental): bolus administration
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Human Milk Oligosaccharides (HMOs) — HMOs will be applied as a neutral-flavoured powder
  Arms: Intervention
Dietary Supplement: Control — will be applied as powder
  Arms: Control

SUMMARY:
Human milk oligosaccharides (HMOs) have been associated with beneficial health outcomes in breastfed infants, therefore they were investigated intensively within recent years. HMOs support the establishment of a "balanced" intestinal microbiome by acting as both a prebiotic and as a specific antimicrobial. In vitro work has demonstrated that HMOs are resistant to hydrolysis by salivary, pancreatic, and brush-border enzymes, as well as to low gastric pH values enzymes. Consequently, HMOs are mostly resistant to digestion and reach the colon unmodified, where they are available for selective utilisation by certain bacteria. Microbial utilisation results in the formation of microbial metabolites, which are associated with local and systemic effects. Simultaneously, HMOs have bacteriostatic effects and directly limit the growth of potential pathogens. Moreover, they serve as antiadhesives, mimicking intestinal epithelial cell surface receptors to which pathogenic microbes attach, thus acting as a decoy receptor. Additionally, it is suggested that HMOs exert effects independent of the microbiome, by modulating cell recognition and cell signalling. These include interactions with immune cells, thereby modulating the development and responses of the immune system, the maturation of the intestinal glycocalyx, and the promotion of neurodevelopment and cognitive functions. A prerequisite for systemic effects is that HMOs are absorbed and can enter the blood circulation, thus making them potentially available at the systemic level. In order to understand the underlying mechanisms for HMO-mediated, microbe-independent effects, information regarding absorption, metabolisation, and excretion is needed and will be investigated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-40 Years
* Non-smoker
* Normal weight (BMI 18.5-25.0 kg/m²)

Exclusion Criteria:

* Impaired insulin sensitivity/glucose tolerance
* Underweight or overweight/obesity
* Regular intake of nutritional supplements
* Alcohol, drug or medication abuse
* Pregnancy and breastfeeding
* Hypo- and hypertension
* Epilepsy
* known hepatitis B, hepatitis C, HIV infection
* Malabsorption and maldigestion syndrome
* Type 1 or type 2 diabetes mellitus
* Other metabolic diseases
* Chronic inflammatory diseases
* Other chronic diseases
* Psychiatric illnesses
* Participation in another study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Absorption of HMOs | through study completion, an average of 1 year
  Concentration of HMOs in blood
Excretion of HMOs | through study completion, an average of 1 year
  Concentration of HMOs in urine

SECONDARY OUTCOMES:
Metabolism | through study completion, an average of 1 year
  Concentration of metabolic markers in blood

CONTACTS AND LOCATIONS:
Locations (1):
- Rheinische Friedrich-Wilhelms Universität Bonn, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No